CLINICAL TRIAL: NCT02616432
Title: Tomosynthesis Mammography Imaging Screening Trial Lead-in
Brief Title: Tomosynthesis Mammographic Imaging Screening Trial
Acronym: TMISTLead-in
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Eastern Cooperative Oncology Group (Network)
Responsible Party: Principal Investigator, Dr. Roberta Jong, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 001-2014b; 410000662 (Other Grant/Funding Number: Canadian Breast Cancer Foundation)
Record Dates: First submitted 2015-11-10; First posted 2015-11-27 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Tomosynthesis; Digital Breast Tomosynthesis (DBT); Breast Imaging; Full-field digital mammography; Breast screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tomosynthesis + FFDM (Experimental): Women enrolled to DBT Arm will undergo manufacturer-defined DBT
  Interventions: Device: Tomosynthesis
- FFDM - Standard of Care for Screening (No Intervention): Women enrolled to the FFDM Arm will undergo bilateral digital mammogram with standard CC and MLO views acquired

INTERVENTIONS:
Device: Tomosynthesis — Three-dimensional imaging of both breasts in standard CC and MLO views
  Arms: Tomosynthesis + FFDM

SUMMARY:
A randomized screening trial to compare the diagnostic accuracy of screening for breast cancer with three-dimensional digital breast tomosynthesis (DBT) plus two-dimensional full-field digital mammography (FFDM) versus FFDM alone.

DETAILED DESCRIPTION:
The Tomosynthesis Mammography Imaging Screening Trial (TMIST) LEAD-IN is being conducted to ensure that all Eastern Cooperative Oncology Group / American College of Radiology Imaging Network (ECOG/ACRIN) TMIST components are properly functional and to provide an opportunity for fine tuning before launching the full TMIST. The accrual target for TMIST LEAD-IN is 6354 participants (one tenth of the projected enrollment target for TMIST) at three lead-in study sites: 1. Sunnybrook Health Sciences Centre in Toronto, 2. Vancouver (under the auspices of the Screening Mammography Programme of British Columbia) and 3. The Ottawa Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic women age 40 and over
* Scheduled for screening mammogram
* Able to tolerate digital breast tomosynthesis and full-field digital mammographic imaging required by protocol
* Willing and able to provide a written informed consent.

Exclusion Criteria:

* Presenting for mammography with symptoms of breast disease
* Have new breast complaints (e.g. lump, nipple discharge)
* Have had a mammogram of both breasts within the last 11 months
* Previous personal history of breast cancer
* Has breast enhancements (e.g. implants or injections)
* Pregnancy or intent to become pregnant.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 3065 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of DBT vs FFDM - AUC under ROC comparison | 3 year follow-up
  To compare the diagnostic accuracy using the area under the curve (AUC) score generated by receiver operator characteristic (ROC) analysis of digital breast tomosynthesis plus full-field digital mammography (DBT) versus full-field digital mammography (FFDM) alone for breast cancer screening. The examinations will be interpreted by local Breast Imaging radiologists. Cancer status will be pathologically confirmed. The women would undergo three consecutive screening rounds in the assigned arm followed by one year of standard of care imaging follow-up.

SECONDARY OUTCOMES:
Recall Rates | 3 year
  To compare the recall rates due to abnormal screening examinations for DBT versus FFDM when used for breast cancer screening.
Interval Cancers | 3 year
  To compare the number of interval cancers missed with DBT versus FFDM use in breast cancer screening.
Prevalence of Breast Cancer Subtypes | 3 year
  To estimate the prevalence of breast cancer subtypes (Luminal A, Luminal B, HER2neu, Basal-like, Claudin-low) by DBT and FFDM, stratified on whether cancers were detected in screening or as interval cancers.
Clinical Characteristics of Cancers | 3 year
  To assess and compare clinical characteristics (e.g. stage, grade, ER, PR, and HER2status) of cancers detected from screening by DBT and FFDM. Approximately 75 genes will be assayed in tumors detected in each arm of the study to evaluate breast cancer molecular subtype.
Reader Studies of variations of DBT vs FFDM - AUC under ROC comparison | 4 year
  To assess different combinations of FFDM, tomosynthesis and synthesized FFDM images in reader studies to assist in determining the optimum balance between radiation exposure and technique. AUC of ROC curves will be used to compare combinations. A panel of radiologists will read the various combinations of images in random order to assess whether tomosynthesis with synthetic 2D images is as accurate as tomosynthesis with FFDM images. The latter will require more radiation exposure.
Biomarker Correlation | 2 year
  Biomarker correlation to characterize disease in the tumor and compare to the tissue immediately adjacent to it.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Jong, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (4):
- Canada (4):
  - X-Ray 505 (Under the BCCA Screening Mammography Program of BC), Vancouver, British Columbia
  - Breast Health Centre at BC Women's Hospital + Health Centre, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
ECOG/ACRIN TMIST will collect all data when accrual starts for that trial.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Immediate
Access Criteria: ECOG/ACRIN Sharing Access policy